CLINICAL TRIAL: NCT05827380
Title: Adaptability Training for Individuals After Stroke
Brief Title: Gait Adaptability Training, Using Augmented Reality, for Individuals in the Chronic Phase After Stroke
Acronym: ATTAINS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sint Maartenskliniek (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL80178.091.21 / 0996
Record Dates: First submitted 2023-02-07; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Patients assigned to the training group will receive a training targeting on gait adaptability using the C-mill. Subjects are asked to stop any other physical therapy program targeting gait, balance or leg function during the training period. Assessments will take place pre- and post-intervention
  Interventions: Behavioral: Gait adaptability training
- Waitlist control group (No Intervention): Patients assigned to the waitlist control group will receive standard care for 5 weeks whereafter they will receive the same training as the training group. Assessments will take place pre-intervention, post-waiting period and post-intervention.

INTERVENTIONS:
Behavioral: Gait adaptability training — During a period of approximately 5 weeks participants will receive 10 one hour training sessions aimed at improving gait adaptability, using the C-mill (an instrumented treadmill with augmented reality). Several aspects of gait adaptability, such as obstacle avoidance, accelerating/decelerating and precision stepping, will be offered.
  Arms: Training group

SUMMARY:
Background: The majority of stroke survivors regain walking ability, however the ability to adapt their gait to meet environmental demands remains impaired. This impaired gait adaptability has a profound impact on activities of daily living and quality of life. Treatment targeting these gait deficiencies is, therefore, critical for allowing safe and independent community ambulation in people with stroke. Rehabilitation programs targeting gait adaptability have gained interest in clinical practice. Besides, the use of augmented and virtual reality in rehabilitation programs becomes more common. Concerning gait adaptability, training programs are developed using the Cmill, an instrumented treadmill with augmented reality. Even though the efficacy of these interventions is limited to small, pilot trials, results are promising. Based on these results we hypothesize that a gait training program using the Cmill will improve gait adaptability and daily-life gait performance in people in the chronic phase after stroke.

Objective: The primary objective of this study is to evaluate the efficacy of a gait training program using an instrumented treadmill with virtual and augmented reality for improving gait adaptability in people in the chronic phase after stroke. A second objective is to identify patient characteristics that predict a more favorable response to training.

Study design: Randomized, waiting-list controlled trial to evaluate gait adaptability training

Study population: 84 stroke patients in the chronic phase after stroke

ELIGIBILITY:
Inclusion Criteria:

* > 6 months after first unilateral supratentorial stroke (chronic phase)
* Able to walk at least 10 minutes independently

Exclusion Criteria:

* Any other neurological or musculoskeletal disease affecting gait or balance (e.g. Parkinson's disease, knee osteoarthritis)
* Contractures or spasticity requiring other treatment (e.g. botulinum toxin treatment) within the duration of the training period.
* Has received multiple training sessions on C-Mill or GRAIL in the past 12 months
* Severe cognitive or visuo-spatial impairments limiting comprehension of instructions or correct perception of the environments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Walking Adaptability Ladder Test (WALT) score | Within 1 week post-intervention
  Measure of gait adaptability. An adapted version for adults of the Walking Adaptability Laddertest for Kids (WAL-K) to assess the ability to flexibly adjust the gait pattern during overground walking. Outcome is based on performance time and foot placement errors measured in seconds where a lower score is a better outcome.
Emory Functional Ambulation Profile (EFAP) score | Within 1 week post-intervention
  Measure of gait adaptability. In this task the participants traverse a standardized 5m obstacle course. Outcome is time to perform the task measured in seconds where a lower score is a better outcome.

SECONDARY OUTCOMES:
Lab-based walking adaptability test | Within 1 week post-intervention
  Measure of gait adaptability. Target stepping task using the Gait Real-time Analysis Interactive Lab (GRAIL) where participant must step on projected stepping stones as accurately as possible. Step width and step length between the stepping stones will vary.
Balance performance | Within 1 week post-intervention
  Measure of gait stability, measured by the margin of stability (meter) and the center of mass excursion (meter), on treadmill walking with perturbations using the Gait Real-time Analysis Interactive Lab (GRAIL).
Balance performance through MiniBESTest | Within 1 week post-intervention
  Measure of balance and gait stability using the Mini Balance Evaluation Systems Test (MiniBESTes). Tasks are scored on a 3-point scale. Outcome is an average score ranging between 0 and 1 where a higher score is a better outcome.
Walking performance | Within 1 week post-intervention
  Measure of walking ability using the 10meter walktest, measured in seconds where a lower score is a better outcome
Balance confidence | Within 1 week post-intervention
  Evaluating balance confidence using the Activity Balance Scale, measured on a 0% - 100% scale, where a higher score is a better outcome
Daily life gait performance as assessed by gait quality | Within 1 week post-intervention
  Measured by inertial measurement units placed on both feet and the lower back. Analysis through cusomized algorythms.
Daily life walking activity assessed by walking time per day | Within 1 week post-intervention
  Average time of walking during the day (minutes) measured in one week using the Activ8.
Health-related quality of life | Within 1 week post-intervention
  Evaluating the disability and health-related quality of life after stroke using the Stroke Impact Scale mobility subscale, measure on a 5-point scale ("could not do at all = 1" - "not difficult at all = 5") where a higher score is a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Weerdesteyn, Prof. dr., Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Ubbergen, Netherlands

REFERENCES:
- [Background] Kuijpers R, Smulders E, Groen BE, Smits-Engelsman BCM, Nijhuis-Van der Sanden MWG, Weerdesteyn V. Reliability and construct validity of the Walking Adaptability Ladder Test for Kids (WAL-K): a new clinical test for measuring walking adaptability in children. Disabil Rehabil. 2022 Apr;44(8):1489-1497. doi: 10.1080/09638288.2020.1802523. Epub 2020 Aug 10. PMID 32776854
- [Background] Tuijtelaars J, Roerdink M, Raijmakers B, Nollet F, Brehm MA. Polio survivors have poorer walking adaptability than healthy individuals. Gait Posture. 2021 Jun;87:143-148. doi: 10.1016/j.gaitpost.2021.04.031. Epub 2021 Apr 21. PMID 33915437
- [Derived] Nieuwelink M, Smulders K, Kamphuis J, Nonnekes J, Keijsers N, Weerdesteyn V. Walking adaptability training for individuals after stroke (ATTAINS): study protocol for a randomized, waiting-list controlled trial. Trials. 2025 Nov 27;26(1):595. doi: 10.1186/s13063-025-09276-w. PMID 41310779
- See also: The project description on the website of the Sint Maartenskliniek (where the study will be performed). — https://www.maartenskliniek.nl/research-innovation/research-innovation-projecten/attains-trainen-van-het-loopaanpassingsvermogen-bij-mensen-na-een-beroerte
- See also: The English description of the project on the website of the Sint Maartenskliniek. — https://www.maartenskliniek.nl/research-innovation-en/research-innovation-projects/attains-gait-adaptability-training-for-people-after-stroke